CLINICAL TRIAL: NCT04443075
Title: Alterations of Gut Microbiome in the Frontline Medical Staff Under the Stress of Fighting Against 2019-nCoV
Brief Title: Alterations of Gut Microbiome in the Frontline Medical Staff Under the Stress
Acronym: AGMFMSS
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2020LSK-022
Record Dates: First submitted 2020-06-03; First posted 2020-06-23 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gut microbiome DNA in faecal samples from included subjects will be extracted and sequnced for the statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exposed group: The exposed group consists of the frontline medical workers who take part in the medical team to support Wuhan.
  Interventions: Device: faecal sample collector
- non-exposed group: This group includs medical workers who didn't join in the medical team to support Wuhan.
  Interventions: Device: faecal sample collector

INTERVENTIONS:
Device: faecal sample collector — The frontline medical workers mainly exposed under the stress of fighting against 2019-nCoV

SUMMARY:
With the outbreak of 2019 novel coronavirus (2019-nCoV), the frontline medical workers faced enormous stress, including a high risk of infection and inadequate protection from contamination, isolation, patients with negative emotions, a lack of contact with their families, and exhaustion, which may cause mental health problems. The investigators plan to collect the faecal samples and clinical assessments from a part of frontline medical workers in three time points to analyse the changing profile of gut microbiome according to outcomes of 16s rRNA sequencing. The samples from the matched health controls will also be sequenced to compare with the exposed group in gut microbiome community.

DETAILED DESCRIPTION:
In December, 2019, a novel coronavirus outbreak of pneumonia emerged in Wuhan, Hubei province, China, and has subsequently spread to more than 30 provinces in China and almost 100 countries in the world. In the fight against the 2019 novel coronavirus (2019-nCoV), medical workers in Wuhan have been facing enormous stress, including a high risk of infection and inadequate protection from contamination, isolation, patients with negative emotions, a lack of contact with their families, and exhaustion. The severe situation is causing mental health problems such as stress, anxiety, depressive symptoms, insomnia, denial, anger, and fear. These mental health problems could also cause posttraumatic stress (PTS) symptoms in a lasting time. A research examining the psychological impact of the 2003 outbreak of severe acute respiratory syndrome on hospital empoyees found that about 10% of the respondents had experienced high leves of PTS symptoms since the SARS outbreak.

Microbiome-gut-brain (MGB) axis has been validated in expanding studies, which means there are bidirectional communication between commensal organisms within the gut and the brain. Gut microbiota may influence brain function through neural, endocrine, and immune pathways. For example, substances produced by the gut microbiota may be absorbed reaching the brain by the blood stream. The brain, in turn, may influence the gut microbiota trough neuronal and endocrine pathways. In recent years, many reseaches support the relevance of microbiota and mental health status. Bercik et al. transplanted microbiota from adult germ-free (GF) BALB/c mice (a high-anxiety mouse strain) into adult GF NIH Swiss mice (a low-anxiety mouse strain), then found the behavioral profile of the donor was evident in the recipient animal, showing that the microbiota can directly affect behavior. Moreover, preclinical studies have shown that stress and emotions, including maternal separation and restraint, heat, and acoustic stress, alters the composition of the gut microbiota, maybe through the release of stress hormones or sympathetic neurotransmitters that influence gut physiology and alter the habitat of the microbiota. In addition, researchers found that stress has the ability to increase intestinal permeability, probably through the involvement of corticotrophin releasing factor and its receptors (CRFR1 and CRFR2), which play a key role in stress-induced gut permeability dysfunction. Increased intestinal permeability provides bacteria an opportunity to translocate across the intestinal mucosa and directly access both the immune and neuronal cells of the enteric nervous system (ENS). Stress also activates the autonomic nervous system, which affects gastric acid, bile, and mucus secretion, as well as gut motility. Gut motility is of particular importance since it is strongly associated with gut microbiota composition and richness. Based on these researches, the gut microbiome increasingly deserve attention to understand psychiatric disorders.

Therefore, the present study aim to collect the faecal samples and clinical assessments from a part of frontline medical workers in three time points to analyse the changing profile of gut microbiome according to outcomes of 16s rRNA sequencing. The samples from the matched health controls will also be sequenced to compare with the exposed group in gut microbiome community.

Methods Study design and sample collection The frontline workers in First Affiliated Hospital of Xi'an Jiaotong University will be included if they conformed with (1) taking part in the medical team to support Wuhan, (2) of 18 to 50 years old, (3) did not take antibiotics within 3 months before sample collection, (4) 17.5<body mass index (BMI)<30. The healthy controls will be selected from the staffs in First Affiliated Hospital who didn't join in the medical team but fulfill the last three conditions above to match with the frontline staffs for age, gender, BMI, and diet. Any participant will be excluded if he/she fulfill the following criteria: (1) have serious cardiovascular disease, blood disease, and endocrine disease, (2) have a history of cancer or its complications, (3) have active gastrointestinal diseases or complications and serious systemic diseases, (4) have history of brain organic diseases or complications and mental retardation, (5) have mental disorders such as mood disorder and anxiety disorders, (6) pregnant or lactating, (7) drink in the past week (liquor>250ml or beer>1bottle) or the previous day (liquor>50ml or beer>50ml). All included persons should provide signed informed consent before sample collection, and the protocol was approved by the Ethics Committee of First Affiliated Hospital of Xi'an Jiaotong University (KYLLSL-2020-043). Faecal samples from each staff should be freshly collected at the hospital and frozen at -80℃ using specified faecal collector.

Clinical assessmant PHQ-15, PHQ-9, GAD-7, PSQI, SCL-90, and IES-R will be used for the assessment of clinical symptoms related to psychiatric disorder for exposed group in three time point and non-exposed group.

DNA extraction and 16S rRNA sequencing The investigators will perform 16S rRNA sequencing for all the collected faecal samples. Briefly, bacterial genomic DNA will be extracted, and the 16S rRNA whole region will be amplified by PCR, and then sequenced.

Statistical analysis The 16S rRNA sequencing data will be analysed using Quantitative Insights Into Microbial Ecology (QIIME). The investigators then use usearch to cluster sequences into taxonomic units (OTUs) at 97% identity and construct the OTU table. Microbial community structure, alpha diversity, and beta diversity will be analysed. LEfSe analysis, and random forest analysis will be used to find the biomarker between different group. Spearman's rank correlation will be used to identify the corrolation between clinical assessments and stress-associated microbiome.

ELIGIBILITY:
Inclusion Criteria:

* taking part in the medical team to support Wuhan
* of 18 to 50 years old
* did not take antibiotics within 3 months before sample collection
* 17.5<body mass index (BMI)<30

Exclusion Criteria:

* have serious cardiovascular disease, blood disease, and endocrine disease
* have a history of cancer or its complications
* have active gastrointestinal diseases or complications and serious systemic diseases
* have history of brain organic diseases or complications and mental retardation
* have mental disorders such as mood disorder and anxiety disorders
* pregnant or lactating
* drink in the past week (liquor>250ml or beer>1bottle) or the previous day (liquor>50ml or beer>50ml)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: They are all medical staff in First Affiliated Hospital of Xi'an Jiaotong University
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Gut microbiome composition of exposed group | immediately after the frontline workers come back to Xi'an
  Gut microbiome composition will be anaylysed using 16S rRNA sequencing.
Gut microbiome composition of exposed group | immediately after the frontline workers isolated for two weeks
  Gut microbiome composition will be anaylysed using 16S rRNA sequencing.
Gut microbiome composition of exposed group | immediately after the frontline workers going back to normal work for one month
  Gut microbiome composition will be anaylysed using 16S rRNA sequencing.
Gut microbiome composition of non-exposed group | During the procedure of collecting faecal samples from exposed group
  Gut microbiome composition will be anaylysed using 16S rRNA sequencing.
The Impact of Event Scale-Revised (IES-R) of exposed group | immediately after the frontline workers come back to Xi'an
  It's a self-report measure assessing subjective distress resulting from a traumatic life event, with a total score of 0-88. Higher score means a worse outcome
The Impact of Event Scale-Revised (IES-R) of exposed group | immediately after the frontline workers isolated for two weeks
  It's a self-report measure assessing subjective distress resulting from a traumatic life event, with a total score of 0-88. Higher score means a worse outcome
The Impact of Event Scale-Revised (IES-R) of exposed group | immediately after the frontline workers going back to normal work for one month
  It's a self-report measure assessing subjective distress resulting from a traumatic life event, with a total score of 0-88. Higher score means a worse outcome
The Impact of Event Scale-Revised (IES-R) of non-exposed group | During the procedure of collecting faecal samples from non-exposed group
  It's a self-report measure assessing subjective distress resulting from a traumatic life event, with a total score of 0-88. Higher score means a worse outcome

SECONDARY OUTCOMES:
The 15-item Patient Health Questionnaire (PHQ-15) of exposed group | immediately after the frontline workers come back to Xi'an
  It's a self-administered measure assessing subjective common mental health with a total score of 0-30. Higher score means a worse outcome.
The 15-item Patient Health Questionnaire (PHQ-15) of exposed group | immediately after the frontline workers isolated for two weeks
  It's a self-administered measure assessing subjective common mental health with a total score of 0-30. Higher score means a worse outcome.
The 15-item Patient Health Questionnaire (PHQ-15) of exposed group | immediately after the frontline workers going back to normal work for one month
  It's a self-administered measure assessing subjective common mental health with a total score of 0-30. Higher score means a worse outcome.
The 15-item Patient Health Questionnaire-15 (PHQ-15) of non-exposed group | During the procedure of collecting faecal samples from non-exposed group
  It's a self-administered measure assessing subjective common mental health with a total score of 0-30. Higher score means a worse outcome.
The 9-item Patient Health Questionnaire (PHQ-9) of exposed group | immediately after the frontline workers come back to Xi'an
  It's a self-report measure widely used for major depression screening with a total score of 0-27. Higher score means a worse outcome.
The 9-item Patient Health Questionnaire (PHQ-9) of exposed group | immediately after the frontline workers isolated for two weeks
  It's a self-report measure widely used for major depression screening with a total score of 0-27. Higher score means a worse outcome.
The 9-item Patient Health Questionnaire (PHQ-9) of exposed group | immediately after the frontline workers going back to normal work for one month
  It's a self-report measure widely used for major depression screening with a total score of 0-27. Higher score means a worse outcome.
The 9-item Patient Health Questionnaire (PHQ-9) of non-exposed group | During the procedure of collecting faecal samples from non-exposed group
  It's a self-report measure widely used for major depression screening with a total score of 0-27. Higher score means a worse outcome.
The 7-item Generalized Anxiety Disorder Scale (GAD-7) of exposed group | immediately after the frontline workers come back to Xi'an
  It is a practical self-report anxiety questionnaire with a total score of 0-21. Higher score means a worse outcome.
The 7-item Generalized Anxiety Disorder Scale (GAD-7) of exposed group | immediately after the frontline workers isolated for two weeks
  It is a practical self-report anxiety questionnaire with a total score of 0-21. Higher score means a worse outcome.
The 7-item Generalized Anxiety Disorder Scale (GAD-7) of exposed group | immediately after the frontline workers going back to normal work for one month
  It is a practical self-report anxiety questionnaire with a total score of 0-21. Higher score means a worse outcome.
The 7-item Generalized Anxiety Disorder Scale (GAD-7) of non-exposed group | During the procedure of collecting faecal samples from non-exposed group
  It is a practical self-report anxiety questionnaire with a total score of 0-21. Higher score means a worse outcome.
The Pittsburgh Sleep Quality Index (PSQI) of exposed group | immediately after the frontline workers come back to Xi'an
  It is a self-report questionnaire that is widely used to assess several dimensions of sleep with a total score of 0-21. Higher score means a worse outcome
The Pittsburgh Sleep Quality Index (PSQI) of exposed group | immediately after the frontline workers isolated for two weeks
  It is a self-report questionnaire that is widely used to assess several dimensions of sleep with a total score of 0-21. Higher score means a worse outcome
The Pittsburgh Sleep Quality Index (PSQI) of exposed group | immediately after the frontline workers going back to normal work for one month
  It is a self-report questionnaire that is widely used to assess several dimensions of sleep with a total score of 0-21. Higher score means a worse outcome
The Pittsburgh Sleep Quality Index (PSQI) of non-exposed group | During the procedure of collecting faecal samples from non-exposed group
  It is a self-report questionnaire that is widely used to assess several dimensions of sleep with a total score of 0-21. Higher score means a worse outcome
The Symptom Check List 90 (SCL-90) of exposed group | immediately after the frontline workers come back to Xi'an
  It is a self-report instrument widely used to measure clinical psychiatric symptoms and mental health status, with a total score of 0-360. Higher means a worse outcome.
The Symptom Check List 90 (SCL-90) of exposed group | immediately after the frontline workers isolated for two weeks
  It is a self-report instrument widely used to measure clinical psychiatric symptoms and mental health status, with a total score of 0-360. Higher means a worse outcome.
The Symptom Check List 90 (SCL-90) of exposed group | immediately after the frontline workers going back to normal work for one month
  It is a self-report instrument widely used to measure clinical psychiatric symptoms and mental health status, with a total score of 0-360. Higher means a worse outcome.
The Symptom Check List 90 (SCL-90) of non-exposed group | During the procedure of collecting faecal samples from non-exposed group
  It is a self-report instrument widely used to measure clinical psychiatric symptoms and mental health status, with a total score of 0-360. Higher means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Xiancang Ma, M.D., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang C, Horby PW, Hayden FG, Gao GF. A novel coronavirus outbreak of global health concern. Lancet. 2020 Feb 15;395(10223):470-473. doi: 10.1016/S0140-6736(20)30185-9. Epub 2020 Jan 24. No abstract available. PMID 31986257
- [Background] Kang L, Li Y, Hu S, Chen M, Yang C, Yang BX, Wang Y, Hu J, Lai J, Ma X, Chen J, Guan L, Wang G, Ma H, Liu Z. The mental health of medical workers in Wuhan, China dealing with the 2019 novel coronavirus. Lancet Psychiatry. 2020 Mar;7(3):e14. doi: 10.1016/S2215-0366(20)30047-X. Epub 2020 Feb 5. No abstract available. PMID 32035030
- [Background] Malan-Muller S, Valles-Colomer M, Raes J, Lowry CA, Seedat S, Hemmings SMJ. The Gut Microbiome and Mental Health: Implications for Anxiety- and Trauma-Related Disorders. OMICS. 2018 Feb;22(2):90-107. doi: 10.1089/omi.2017.0077. Epub 2017 Aug 2. PMID 28767318
- [Background] Foster JA, McVey Neufeld KA. Gut-brain axis: how the microbiome influences anxiety and depression. Trends Neurosci. 2013 May;36(5):305-12. doi: 10.1016/j.tins.2013.01.005. Epub 2013 Feb 4. PMID 23384445
- [Background] Wu P, Fang Y, Guan Z, Fan B, Kong J, Yao Z, Liu X, Fuller CJ, Susser E, Lu J, Hoven CW. The psychological impact of the SARS epidemic on hospital employees in China: exposure, risk perception, and altruistic acceptance of risk. Can J Psychiatry. 2009 May;54(5):302-11. doi: 10.1177/070674370905400504. PMID 19497162
- [Background] Rieder R, Wisniewski PJ, Alderman BL, Campbell SC. Microbes and mental health: A review. Brain Behav Immun. 2017 Nov;66:9-17. doi: 10.1016/j.bbi.2017.01.016. Epub 2017 Jan 25. PMID 28131791